CLINICAL TRIAL: NCT03597867
Title: Vitreous pge2 Level Changes After Topical Administration of Diclofenac 0.1%, Nepafenac 0.3%, Indomethacin 0.5% and Bromfenac 0.09% in Vitrectomy Patients
Brief Title: PGE2 Levels in Patient Treated With NSAIDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Marco Rocco Pastore, Principal Investigator, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02/2017
Record Dates: First submitted 2018-07-11; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Ocular Inflammation
Keywords: vitreoretinal surgery; epiretinal membrane; macular hole; non steroidal antinflammatory drugs; prostaglandin E2
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations | interventions — nepafenac; Indomethacin; bromfenac; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo using single-use vials of hyaluronic acid 0.2% preservative-free lubricating tear drops three days before surgery.
  Interventions: Other: Placebo
- Dicloftil (Experimental): Diclofenac Na 0.1% Oph Soln, "Dicloftil®", NSAID eyedrops administered three days before surgery
  Interventions: Drug: Dicloftil
- Nevanac (Experimental): Nepafenac 0.3% Ophthalmic Suspension, "Nevanac 3mg/ml®", NSAID eyedrops administered three days before surgery
  Interventions: Drug: Nevanac
- Indom (Experimental): Indomethacin 5 MG/ML Ophthalmic Suspension, "Indom ®", NSAID eyedrops administered three days before surgery
  Interventions: Drug: Indom
- Yellox (Experimental): Bromfenac 0.09 % Ophthalmic Solution, "Yellox®", NSAID eyedrops administered three days before surgery
  Interventions: Drug: Yellox

INTERVENTIONS:
Other: Placebo — Artificial tears for 3 days preoperatively
  Other Names: Tears
  Arms: Placebo
Drug: Dicloftil — Dosing of drug 3 days prior to surgery
  Other Names: Diclofenac Na 0.1% Oph Soln
  Arms: Dicloftil
Drug: Nevanac — Dosing of drug 3 days prior to surgery
  Other Names: Nepafenac 0.3% Ophthalmic Suspension
  Arms: Nevanac
Drug: Indom — Dosing of drug 3 days prior to surgery
  Other Names: Indomethacin 5 MG/ML Ophthalmic Suspension
  Arms: Indom
Drug: Yellox — Dosing of drug 3 days prior to surgery
  Other Names: Bromfenac 0.09 % Ophthalmic Solution
  Arms: Yellox

SUMMARY:
The aim of this study is to determine vitreous levels of nonsteroidal antinflammatory drugs (NSAIDs) and prostaglandinE2 (PGE2) in eyes scheduled for vitrectomy.

All patients received the study drugs for 3 days before surgery. 0.5 to 1.0 mL of undiluted vitreous was removed using the vitreous cutter positioned in the midvitreous cavity. Samples were immediately frozen and stored at -80°C until analysis.

Sample analyses were performed using an high-performance liquid chromatography system. The lower limit of quantitation was 0.8 ng/mL.

PGE2 levels were analyzed using the Prostaglandin E2 Monoclonal EIA Kit (Cayman Chemical Company) according to the manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* epiretinal membrane or full thickness macular hole scheduled for vitrectomy

Exclusion Criteria:

* vitreous hemorrhage
* diabetes
* glaucoma
* concurrent retinovascular disease
* previous ocular inflammation
* previous ocular surgery
* history of ocular trauma
* previuos intravitreal injections
* concomitant intake of topical or systemic NSAIDs or corticosteroid therapy

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
Vitreous NSAIDs and PGE2 levels | 3 days after topical NSAID administration

CONTACTS AND LOCATIONS:
Overall Officials: Marco R Pastore, MD, Principal Investigator — Eye Clinic, Departement of Medical Surgical Sciences and Health, University of Trieste Trieste, TS, 34129, Italy
Locations (1):
- Eye Clinic, Departement of Medical Surgical Sciences and Health, University of Trieste, Trieste, TS, Italy

IPD SHARING:
Plan to Share IPD: No